CLINICAL TRIAL: NCT04047680
Title: Evolution of Estimated Glomerular Filtration Rate in Chronic Hepatitis C Patients Receiving Sofosbuvir-based or Sofosbuvir-free Direct Acting Antivirals
Brief Title: eGFR Evolution in HCV Patients Receiving SOF-based or SOF-free DAAs
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201509009RINB
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C; Renal Disease; Viral Hepatitis C
Keywords: Viral hepatitis C; Glomerular filtration rate; Direct acting antiviral agent; Sofosbuvir
MeSH Terms: conditions — Hepatitis C; Kidney Diseases | interventions — sofosbuvir-velpatasvir drug combination; ledipasvir, sofosbuvir drug combination; Sofosbuvir; ombitasvir; elbasvir-grazoprevir drug combination; glecaprevir and pibrentasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SOF-based DAAs: Patients receiving sofosbuvir (SOF)-based direct acting antiviral agents (DAAs) for 12 weeks
  Interventions: Drug: Sofosbuvir / Velpatasvir Oral Tablet; Drug: Sofosbuvir and Ledipasvir; Drug: Sofosbuvir Tablets
- SOF-free DAAs: Patients receiving sofosbuvir (SOF)-free direct acting antiviral agents (DAAs) for 12 weeks
  Interventions: Drug: Ombitasvir/paritaprevir/ritonavir; Drug: Elbasvir / Grazoprevir Oral Tablet; Drug: Glecaprevir and Pibrentasvir

INTERVENTIONS:
Drug: Sofosbuvir / Velpatasvir Oral Tablet — Sofosbuvir/velpatasvir for 12 weeks
  Other Names: Epclusa
  Groups: SOF-based DAAs
Drug: Sofosbuvir and Ledipasvir — Sofosbuvir and ledipasvir for 12 weeks
  Other Names: Harvoni
  Groups: SOF-based DAAs
Drug: Sofosbuvir Tablets — Sofosbuvir plus ribavirin (RBV) or daclatasvir (DCV) for 12 weeks
  Other Names: Solvadi
  Groups: SOF-based DAAs
Drug: Ombitasvir/paritaprevir/ritonavir — Ombitasvir/paritaprevir/ritonavir for 12 weeks
  Other Names: Viekirax/exviera
  Groups: SOF-free DAAs
Drug: Elbasvir / Grazoprevir Oral Tablet — Elbasvir/grazoprevir for 12 weeks
  Other Names: Zepatier
  Groups: SOF-free DAAs
Drug: Glecaprevir and Pibrentasvir — Glecaprevir/pibrentasvir for 12 weeks
  Other Names: Maviret
  Groups: SOF-free DAAs

SUMMARY:
Data regarding the nephrotoxicity of sofosbuvir (SOF) remain controversial. The investigators compared the changes of estimated glomerular filtration rate (eGFR) in patients with chronic hepatitis C virus (HCV) infection receiving SOF-based or SOF-free direct acting antivirals (DAAs).

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is a major health problem that affects 71 million people worldwide. Patients with chronic HCV infection may present with various hepatic and extrahepatic manifestations which lead to substantial morbidity and mortality. In contrast, the long-term health outcome improves following successful HCV eradication by antiviral therapies.

Owing to the excellent efficacy and safety as well as the short treatment duration, the use of interferon (IFN)-free direct acting antivirals (DAAs) has become the standard-of-care for managing HCV. Sofosbuvir (SOF) is a pyrimidine nucleotide analogue which acts as the HCV ribonucleic acid (RNA) chain terminator by inhibiting HCV non-structural protein 5B (NS5B) RNA-dependent RNA polymerase following intrahepatic activation to uridine triphosphate form. Dephosphorylation results in the formation of inactive metabolite (GS-331007) that undergoes extensive renal excretion. Clinically, SOF is administered once-daily with pangenotypic potency, well tolerability and a high genetic barrier to drug resistance. Furthermore, SOF can be used in combination with NS3/4A protease inhibitors (PIs), NS5A inhibitors, and/or ribavirin (RBV) to achieve high rates of sustained virologic response (SVR). Therefore, applying SOF-based DAAs for HCV is welcome to most treating physicians.

Following the widespread use of SOF-based DAAs for treating HCV in different populations, a large-scale real-world HCV-TARGET study enrolling 1,789 patients indicated that patients with a baseline eGFR ≤ 45 mL/min/1.73m2 were associated with a higher risk of worsening renal function than those with a baseline eGFR > 45 mL/min/1.73m2 following SOF-based DAAs. Moreover, three retrospective studies showed that SOF-based DAAs negatively affected the on-treatment and off-therapy eGFR. On the contrary, other studies showed that the use of SOF-based DAAs did not worsen the eGFR. Because most studies were retrospective in nature without protocol-defined time point for eGFR assessment or patient election, and did not enroll patients receiving SOF-free DAAs as the controls, the investigators thus conducted a prospective study to evaluate the evolution of eGFR in patients with chronic HCV infection receiving SOF-based or SOF-free DAAs.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV patients receiving SOF-based or SOF-free DAAs for 12 weeks

Exclusion Criteria:

* Decompensated cirrhosis (Child-Pugh B or C)
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2
* Active hepatocellular carcinoma (HCC)
* Organ transplantation
* Hepatitis B virus (HBV) co-infection
* Human immunodeficiency virus (HIV) co-infection
* Not received off-therapy follow-up till week 24

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C virus-infected patients with compensated liver diseases and baseline eGFR of 30 mL/min/1.73m2 or more, who received SOF-based or SOF-free DAAs for 12 weeks, and who received off-therapy follow-up until week 24
Sampling Method: Non-Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Slope differences of eGFR | Baseline to off-therapy week 24
  Slope differences of eGFR between SOF-based and SOF-free DAAs

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Horng Kao, PhD, Study Director — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu CH, Lee MH, Lin JW, Liu CJ, Su TH, Tseng TC, Chen PJ, Chen DS, Kao JH. Evolution of eGFR in chronic HCV patients receiving sofosbuvir-based or sofosbuvir-free direct-acting antivirals. J Hepatol. 2020 May;72(5):839-846. doi: 10.1016/j.jhep.2019.11.014. Epub 2019 Nov 29. PMID 31790766